CLINICAL TRIAL: NCT01154712
Title: Deep Low-Frequency Repetitive Transcranial Magnetic Stimulation for Cessation of Pathological Gambling
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: Dr. Oded Rosenberg, Beer Ya'acov mental health institue
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 244
Record Dates: First submitted 2010-06-30; First posted 2010-07-01 (Estimated); Last update posted 2010-07-14 (Estimated); Status verified 2010-01

CONDITIONS: Pathological Gambling
Keywords: Gambling; Deep TMS; addiction; Brain stimulation
MeSH Terms: conditions — Gambling; Behavior, Addictive

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Real Deep TMS (Active Comparator): Stimulation parameters : Dorso lateral prefrontal cortex,1HZ,600 pulses per session,15 sessions
  Interventions: Device: Real Deep TMS
- Sham Deep TMS (Sham Comparator): Stimulation parameters : Dorso lateral prefrontal cortex,1HZ,600 pulses per session,15 sessions
  Interventions: Device: Sham Deep TMS

INTERVENTIONS:
Device: Real Deep TMS — Stimulation parameters : Dorso lateral prefrontal cortex,1HZ,600 pulses per session,15 sessions
  Arms: Real Deep TMS
Device: Sham Deep TMS — Stimulation parameters : Dorso lateral prefrontal cortex,1HZ,600 pulses per session,15 sessions
  Arms: Sham Deep TMS

SUMMARY:
Pathological gambling (PG) is characterized by a persistent pattern of continued gambling behavior despite its adverse consequences. PG is a chronic, progressive, male-dominated disorder, which has a prevalence of 1% to 3.4% among US adults. Deep transcranial magnetic stimulation (TMS) is a novel neuro-stimulation method capable of inhibiting neuronal activity when given in low frequency. The hypothesis of this study is that , Pathological gambling will be ameliorated if low frequency magnetic field using Brainsway H1 coil will be applied to the left dorso-lateral prefrontal cortex of these patients.

DETAILED DESCRIPTION:
Deep Low-Frequency Repetitive Transcranial Magnetic Stimulation for cessation of pathological gambling

Introduction:

Pathological gambling (PG) is characterized by a persistent pattern of continued gambling behavior despite its adverse consequences. PG is a chronic, progressive, male-dominated disorder, which has a prevalence of 1% to 3.4% among US adults. Typically, the patient's life becomes dominated by the gambling behavior leading to overwhelming financial burdens, an inability to maintain a career, and to the eventual disintegration of family relationships. The enormous personal and social consequences of this disorder include a high rate of suicide attempts, legal problems, and criminal behavior [R1].

Several theoretical models of drug addiction have suggested that addiction is related to abnormal activity in the ventromedial prefrontal cortex system, which is necessary for inhibiting both the craving for immediate reward and excitement-seeking behavior [ref2]. Neuropsychological studies of pathological gamblers [ref 3to9 ref2 ref10] have demonstrated that pathological gamblers have deficits in the frontal lobe/reward system leading investigators to hypothesize that impairment of executive function may play an important role in the etiology of pathological gambling.

Drawing from the field of drug dependence, it has been speculated that the underlying pathology in pathological gambling is a reduction in the sensitivity of the reward system. Reuter et al studied pathological gamblers and controls during a guessing game using functional magnetic resonance imaging and observed a reduction of ventral striatal and ventromedial prefrontal activation in the pathological gamblers that was negatively correlated with gambling severity, linking hypo-activation of these areas to disease severity [ ref11]. Studies in the field of addiction have shown that prefrontal regulation of behavior is reduced in basal conditions, thereby contributing to the reduced salience of non-drug motivational stimuli and reduced decision-making ability. However, when stimuli predicting drug availability are presented, there is profound activation of the prefrontal cortex and glutamatergic drive to the nucleus accumbens [ref12].

Potenza et al in a functional magnetic resonance imaging study demonstrated that male pathological gamblers showed relatively reduced activity in the frontal and orbitofrontal cortex, caudate and basal ganglia and thalamus as compared to controls when presented with visual gambling cues [ref13].Recent neurobehavioral studies have demonstrated poor performance on tests of executive function in pathological gamblers suggesting that the financial risk-taking behavior seen in PG may be associated with both dorsolateral prefrontal and orbitofrontal cortex dysfunction [ref 14-17].Neuropsychological studies of PGs have demonstrated that PGs have deficits in the frontal lobe/reward system [ref18 ref10].Patients with pathological gambling demonstrated greater decreases in binding potential in the ventral striatum during gambling (13.9%) than control patients (8.1%), likely reflecting greater dopaminergic release. Ventral striatal bindings at baseline during control task were also lower in patients with pathological gambling [ref19].

Reductions in right prefrontal activity during decision-making appear to be modulated by the presence of gambling problems and may reflect impaired working memory, stimulus reward valuation, or cue reactivity in substance dependent individuals [ref20].

PG is related to response perseveration and diminished reward and punishment sensitivity as indicated by hypoactivation of the ventrolateral prefrontal cortex when money is gained and lost. Moreover, intact planning abilities and normal dorsal frontostriatal responsiveness indicate that this deficit is not due to impaired executive functioning. Response perseveration and ventral prefrontal hypo-responsiveness to monetary loss may be markers for maladaptive behavior seen in chemical and non-chemical addictions [ref21].

In one study, subjects and 10 matched healthy control subjects underwent fMRI during visual presentations of gambling-related video alternating with video of nature scenes. Pathological gambling subjects and control subjects exhibited overlap in areas of brain activity in response to the visual gambling cues; however, compared with control subjects, PG subjects exhibited significantly greater activity in the right dorsolateral prefrontal cortex (DLPFC), including the inferior and medial frontal gyri, the right parahippocampal gyrus, and left occipital cortex, including the fusiform gyrus [R22].

It has been reported that High-frequency (20-Hz) rTMS of left dorsolateral prefrontal cortex can reduce cigarette smoking significantly [ref23].In another study, found that multiple high-frequency rTMS of the DLPFC can attenuate nicotine craving [ref 24].Regarding cocaine addiction treatment with TMS, it has been shown that one session of 10Hz rTMS over right, but not left, DLPFC transiently reduces craving in cocaine dependent individuals [ref25].Politi et al. conducted a study including thirty-six subjects fulfilling DSM-IV criteria for cocaine dependence. Subjects were treated with 20 trains of TMS applied to the left prefrontal cortex in frequency of 15 Hz and intensity of 100% of the motor threshold. Repeated measures analyses of variance showed that cocaine craving were gradually reduced during sessions of TMS [ref26].

Hypothesis Assuming substance addiction and pathological gambling share similar patho-physiology and considering the evidence that transcranial magnetic stimulation of left dorsolateral prefrontal cortex can ameliorate addiction in both smoking [ ref23 ] and cocaine[ ref26 ] we hypothesize that transcranial magnetic stimulation may also reduce gambling "craving" in pathological gamblers.

H-coil placed over the frontal cortex exerts a significant effect over the entire ipsilateral cortical hemisphere, but significantly less over the contralateral hemisphere [ref27].Thus, the H-coil placed over the DLPFC is hypothesized to exert a direct and more consistent effect on cortical and subcortical regions such as the anterior cingulate and nucleus accumbens (ventral striatum), compared to the figure-8 coil. Because these regions are considered to play a role in drug craving and addiction, rTMS applied with the H-coil may be more effective in reducing drug craving than rTMS applied with the standard figure-8 coil.

Deep TMS:

Deep TMS is currently being evaluated as a treatment option in major depression. It has been shown to be a safe procedure [ref28, ref29]. The innovative design of Brainsway H-Coils is intended to generate sufficient magnetic field strength to stimulate neurons deep inside the brain mass without posing a hazard. This forms the basis of the Brainsway H-Coil used in their deep rTMS device. The coils are designed to maximize the electrical field deep in the brain by the summation of separate fields projected into the skull from several points around its periphery. The device also minimizes the accumulation of electrical charge on the surface of the brain, which can give rise to an electrostatic field that might reduce the magnitude of the induced electric field both at the surface and inside, and reduce the depth penetration of the induced electric field [ref30]. The unique shape of the device's base includes wire coils containing several wire strips, set tangentially to the scalp's surface. Each set of strips is connected in series and contains current flowing in the same direction, therefore generating a field that extends into the brain in a specified orientation from each location along the scalp. Computerized theoretical calculations were made in order to optimize the coil design for maximizing the percentage of stimulation in depth relative to the cortical regions. These, in conjunction with tests performed in a phantom model, [ref 30, ref28, ref27] demonstrated the ability to stimulate, by means of the H-Coil, deep brain regions. It may be assumed then that the activation of deep brain regions and their interconnecting fibers may serve as a new approach in treating neuropsychiatry illnesses with prominent advantage over the standard coil, unable to affect regions as deep as the H-Coil. Deep TMS could be more effective than rTMS due to its deeper penetration into brain tissues [ref28]. The deeper penetration should produce greater action on nerve fibers connecting the prefrontal cortex to the limbic system.

In a randomized controlled study of deep transcranial magnetic stimulation conducted in Israel, 32 healthy volunteers (9 of which were tested for H1 coil presented in this report) were evaluated for possible cognitive impairment. Cognitive evaluation was conducted using the Cambridge Neuropsychological Test Automated Battery (CANTAB), which is sensitive to cognitive changes caused by a wide range of Central Nervous System disorders and medication side-effects. No deterioration in cognitive functions was found, except for a transient short-term effect of the H1-coil on spatial recognition memory on the first day of rTMS (but not in the following treatment days). Questionnaires conducted for emotional or mood alterations, showed no significant changes except for reports on 'detachment' experienced by subjects treated with the H1-coil.In addition, stimulation with the novel H-coils was found to be well tolerated, with no adverse physical or neurological outcomes [ref29].

Contraindications to deep TMS are essentially the same as those for rTMS. Absolute contraindications include history of any metal object in the head, known history of any metallic particles in the eye, implanted cardiac pacemaker or any intra-cardiac lines, implanted neurostimulators, surgical clips or any medical pumps, history of cochlear implants and a history of seizure or heat convulsion. Relative contraindications include epilepsy or seizure in first degree relatives, history of head injury; frequent or severe headaches, migraines; hearing loss; drug abuse or alcoholism, pregnancy or not using a reliable method of birth control and systemic and metabolic disorders.

Methods:

40 patients aged 18-65 years, diagnosed as suffering from pathological gambling according to DSM-IV-TR will be recruited from outpatient treatment programs at the Beer Yaacov Mental Health Center. Within 3 days prior to the first treatment session patients will be assessed by a rater blind to real /sham treatment with the following measures:

1. SCID -version 2
2. Hamilton Depression 24 items
3. Hamilton Anxiety
4. Y-BOCS
5. SOGS (South Oaks Gambling Screen)
6. DAGS (Dannon Ainhold Gambling Scale)
7. VAS (visual analogue scale)
8. CGI-I
9. Social Adaptation Scale (SAS)
10. Complete battery of Neurocognitive tests

Following preliminary assessment, patients will be equally and randomly divided to 2 study arms as described below:

Real TMS Sham TMS Gambling photos \ videos 20 Patients 20 Patients

Real TMS will be given to the Dorso-lateral prefrontal cortex with the following parameters :

* Frequency: 1HZ
* Total number of stimulations per session: 600
* Motor threshold percentage: 120%
* Total duration of treatment session (minutes): 10
* Total number of treatment sessions: 15

Deep TMS coil used in this study will be the H-ADD coil (Please see investigator's brochure).

Patients will undergo 5 courses per week during 3 weeks.

Evaluations (Including the Neurocognitive tests) will be performed 24 hours after the 15th session and again 1 week after the last session and 1 month after the last session.

ELIGIBILITY:
Inclusion Criteria:

* Pathological gambling according to Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition, Text Revision (DSM-IV-TR)

Exclusion Criteria:

* History of a primary major psychiatric or cognitive disorder according to DSM IV apart from Pathological gambling.
* Current alcohol or other substance abuse or dependence.
* Alcohol or other substance abuse or dependence during the last 12 months before recruitment.
* History of or evidence of significant brain malformation or neoplasm, head injury, cerebral vascular events, neurodegenerative disorder affecting the brain or prior brain surgery.
* Significant neurological co-morbidity.
* psychiatric co-morbidity.
* psychotropic medications.
* Severe somatic co morbidity.
* Cardiac pace makers, other electronic implants, intracranial metallic particles.
* History of seizures or epileptiform activity.
* Pregnancy and lactation.
* Patients who cannot communicate reliably with the investigator or who are not likely to cope with the requirements of the experiment.
* Patients unwilling or unable to give written informed consent.
* Patients with a high risk for severe violence or suicidality as assessed during the screening interview.
* Participation in a clinical trial within the last 30 days before the beginning of this clinical trial or similar participation in another clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-06; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
SOGS (South Oaks Gambling Screen) | 45 days
  The South Oaks Gambling Screen is a 20-item questionnaire based on Diagnostic and Statistical Manual of Mental Disorders, Third Edition (DSM-III) criteria for pathological gambling.
Dannon Ainhold Gambling Scale | 45 days
  A scale for assessment of pathological gambling
visual analogue scale | 45 Days
  An instrument for assessment of desire to indulge in gambling

SECONDARY OUTCOMES:
Hamilton Depression 24 items | 45 Days
  Depression assessment scale
Hamilton Anxiety scale | 45 days
  Anxiety assessment scale
Yale-Brown Obsessive Compulsive Scale (Y-BOCS) | 45 days
  A scale for assessment of compulsions and obsessions
Clinical Global Impression Improvement (CGI-I) | 45 days
  A scale for assessment of global clinical improvement
Social Adaptational Scale(SAS) | 45 days
  A scale for assessment of Social Adaptation

CONTACTS AND LOCATIONS:
Overall Officials: Oded Rosenberg, MD, Study Chair — Beer Yaakov Mental Health Center; Pinhas Dannon, MD, Principal Investigator — Beer Yaakov Mental Health Center
Locations (1):
- Beer Yaakov Mental Health Center, Beer Yaakov, Hashfela, Israel